CLINICAL TRIAL: NCT03636347
Title: A Phase 2, Proof-of-concept, Multicentre, Double-blind, Randomised, Dose-ascending, Sequential Group, Placebo-controlled Study to Evaluate the Mechanistic Effect, Safety, and Tolerability of 12 Weeks Twice Daily Oral Administration of Alvelestat (MPH966) in Participants With Alpha-1 Antitrypsin Deficiency.
Brief Title: A 12-week Study Treating Participants Who Have alpha1-antitrypsin-related COPD With Alvelestat (MPH966) or Placebo.
Acronym: ASTRAEUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mereo BioPharma (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MPH966-2-01; 2018-001309-95 (EudraCT Number)
Record Dates: First submitted 2018-06-20; First posted 2018-08-17 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Alpha 1-Antitrypsin Deficiency; Emphysema; COPD
Keywords: PiZZ or Null; Neutrophil elastase inhibitor; Alpha-1; Alvelestat; AZD9668; MPH966; Rare variant genotype; Astraeus; AATD; Alpha 1-Antitrypsin Deficiency; Lung Disease
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Emphysema; Pulmonary Disease, Chronic Obstructive; Lung Diseases

STUDY DESIGN:
Intervention Model Description: placebo-controlled, dose ascending, sequential group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo oral tablet (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet
- Alvelestat oral tablet - dose 1 (Active Comparator): MPH966
  Interventions: Drug: Alvelestat oral tablet - dose 1
- Alvelestat oral tablet - dose 2 (Active Comparator): MPH966
  Interventions: Drug: Alvelestat oral tablet - dose 2

INTERVENTIONS:
Drug: Placebo Oral Tablet — twice daily administration
  Arms: Placebo oral tablet
Drug: Alvelestat oral tablet - dose 1 — twice daily administration
  Other Names: MPH966
  Arms: Alvelestat oral tablet - dose 1
Drug: Alvelestat oral tablet - dose 2 — twice daily administration
  Other Names: MPH966
  Arms: Alvelestat oral tablet - dose 2

SUMMARY:
The purpose of this study is to investigate the effect of alvelestat (an oral neutrophil elastase inhibitor) on blood and sputum biomarkers in patients with PiZZ, null or rare variant phenotype/genotype alpha-1 anti-trypsin deficient lung disease. Change in a number of different blood and sputum biomarkers related to lung damage, inflammation and elastase activity will be measured over a 12 week period. The effect on lung function and respiratory symptoms will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of alpha-1-anti-trypsin deficiency and a PiZZ, null or other rare geno/phenotype and serum anti-alpha1 antitrypsin levels of less than 11uM
* FEV1 ≥20% predicted
* Computerised tomography (CT) scan evidence of emphysema
* Non-smokers

Exclusion Criteria:

* Primary diagnosis of bronchiectasis
* An ongoing acute exacerbation of the underlying lung disease
* Underlying liver disease or abnormal liver function tests
* Previous augmentation therapy within 6 months of dosing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline on blood biomarkers of neutrophil elastase activity compared to baseline and placebo | 12 weeks
  Within-individual change from baseline up to end of treatment in:
  * Blood neutrophil elastase activity
  * Blood Aα-Val 360 levels
  * Plasma desmosine/isodesmosine levels

SECONDARY OUTCOMES:
Change from baseline on other blood biomarkers of neutrophil elastase activity | 12 weeks
  Frequency of neutrophil elastase levels below the limit of detection from baseline to end of treatment

OTHER OUTCOMES:
Change from baseline in St. George's Respiratory Questionnaire (SGRQ-C) to end of treatment | 12 weeks
  Total score
Change from baseline in pulmonary function | 12 weeks
  Change from baseline in forced expiratory volume in 1 second (FEV1)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Stockley, Prof., Principal Investigator — University of Birmingham
Locations (26):
- United States (4):
  - University of Alabama, Birmingham (UAB), Birmingham, Alabama
  - UCLA Medical Center, Los Angeles, California
  - UC Davis Medical Centre, Sacramento, California
  - PMG Research of Wilmington, Wilmington, North Carolina
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Canada (4):
  - The University Lung Clinic, Edmonton, Alberta
  - Centre for Heart Lung Innovation, St Pauls Hospital, Vancouver, British Columbia
  - Inspiration Research Ltd, Toronto, Ontario
  - University of Saskatchewan Royal University Hospital, Saskatoon, Saskatchewan
- Denmark (3):
  - Aarhus Universitetshospital, Aarhus
  - Gentofte Hospital, Hellerup
  - Synddansk Universitet (SDU) - Odense University, Odense
- Instytut Gruzilicy Chorob Pluc, Warsaw, Poland
- Spain (2):
  - Hospital Univ Clinico San Carlos, Madrid
  - Hospital Sierrallana, Torrelavega
- Sweden (2):
  - CTC Gothia Forum Sahlgrenska University Hospital, Gothenburg
  - Lund University Hospital, Lund
- United Kingdom (8):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Cambridge University Hospitals Foundation NHS Trust, Cambridge
  - University Hospital Coventry and Warwickshire, Coventry
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Devon and Exeter NHS Trust, Exeter
  - University Hospitals of Leicester NHS Trust, Leicester
  - Royal Brompton Hospital, London
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No